CLINICAL TRIAL: NCT02397395
Title: A Phase 2, Open-label, Single-arm Study to Investigate the Efficacy, Safety, Tolerability and Pharmacokinetics of 12 Weeks Treatment With Simeprevir and Daclatasvir in Subjects With Chronic Hepatitis C Virus Genotype 1b or 4 Infection and Either Severe Renal Impairment or End-stage Renal Disease on Hemodialysis.
Brief Title: An Efficacy, Safety, Tolerability and Pharmacokinetics Study of 12 Weeks Treatment With Simeprevir and Daclatasvir in Participants With Chronic Hepatitis C Virus Genotype 1b or 4 Infection and Either Severe Renal Impairment or End-stage Renal Disease on Hemodialysis.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial has been cancelled due to availability of new therapeutic options for patient population
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR106396; TMC435HPC2018 (Other: Janssen R&D Ireland); 2014-004250-34 (EudraCT Number)
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Renal Impairment; End-stage Renal Disease
Keywords: Renal Impairment; End-stage Renal Disease; Simeprevir; Daclatasvir
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic | interventions — Simeprevir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Simeprevir Co-administered with Daclatasvir (Experimental): All participants will receive Simeprevir (SMV) 150 milligram (mg) capsule co-administered with Daclatasvir (DCV) 60 mg tablet, orally, once daily for a duration of 12 weeks. Participants should take the study drugs (SMV and DCV together) orally and once daily with food.
  Interventions: Drug: Simeprevir (SMV) 150 mg; Drug: Daclatasvir (DCV) 60 mg

INTERVENTIONS:
Drug: Simeprevir (SMV) 150 mg — Simeprevir (SMV) 150 milligram (mg) capsule orally, once daily for a duration of 12 weeks.
Drug: Daclatasvir (DCV) 60 mg — Daclatasvir (DCV) 60 mg tablet, orally, once daily for a duration of 12 weeks.

SUMMARY:
The purpose of this study is to evaluate the percentage of participants with sustained virologic response 12 weeks after the actual end of study treatment (SVR12)

DETAILED DESCRIPTION:
This is a Phase 2, open-label (identity of study drug will be known to volunteer and study staff), single-arm, multicenter (when more than one hospital work on a medical research study) study to evaluate the efficacy, safety, tolerability and pharmacokinetics of 12 weeks treatment with Simeprevir (SMV) and Daclatasvir (DCV) in participants with chronic Hepatitis C Virus (HCV) genotype 1b or 4 infection and either severe renal impairment or End-stage Renal Disease on hemodialysis. The study consists of a Screening Phase of 4 weeks, an Open-label Treatment Phase of 12 weeks, and a post-Treatment Follow-up Phase of 24 weeks. The total study duration for each participant will be approximately 40 weeks. All participants will receive a treatment regimen consisting of SMV 150 mg and DCV 60 mg co-administered once daily for a total treatment duration of 12 weeks. Participants who experience inadequate virologic response at Week 8 (defined as confirmed HCV RNA greater than or equal to [>=] lower limit of quantification [LLOQ]) or viral breakthrough at any on-treatment visit (defined as confirmed increase in HCV RNA of >1 log base 10 from nadir, or confirmed HCV RNA >100 International unit per milliliter [IU/mL] in participants whose HCV RNA had previously been <LLOQ while on treatment) should discontinue all study drugs. Participants will be primarily evaluated for sustained virologic response 12 weeks after the actual end of study treatment (SVR12). Participants' safety will be evaluated throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, between 18 and 70 years of age, inclusive, at screening
* Hepatitis C Virus (HCV genotype): HCV genotype 1b or 4 (determined at screening)
* Plasma HCV RNA: Greater than (>) 10,000 international unit per milliliter (IU/mL) (determined at screening)
* HCV disease status: FibroScan less than (<) 14.5 kilopascal (kPa), performed within 3 months prior to screening, or between screening and baseline (Day 1), and no history or signs or symptoms of decompensated liver disease. In participants with FibroScan >12.5 kPa, absence of findings suspicious for hepatocellular carcinoma documented by an abdominal ultrasound, performed within 3 months prior to screening, or between screening and baseline (Day 1)
* HCV treatment history: HCV treatment-naive participants, defined as never having received HCV treatment with any approved or investigational drug (including vaccines); OR HCV treatment-experienced, defined as having received previous HCV treatment with any (pegylated) interferon ([Peg]IFN)-based drug regimen (with or without ribavirin [RBV] and not including a direct-acting antiviral agent [DAA]). Last dose in this previous HCV treatment course should have occurred at least 2 months prior to screening

Exclusion Criteria:

* Infection/co-infection: HCV genotype other than 1b or 4, Human immunodeficiency virus type 1 or 2
* Liver disease of non-HCV etiology: Any evidence of liver disease of non-HCV etiology. This includes, but is not limited to, acute hepatitis A, hepatitis B (hepatitis B surface antigen positive), drug- or alcohol-related liver disease, autoimmune hepatitis, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, non-alcoholic steatohepatitis, primary biliary cirrhosis, or any other non-HCV liver disease considered clinically significant by the investigator
* Hepatic decompensation: History or evidence of clinical hepatic decompensation (presence of ascites, bleeding varices or hepatic encephalopathy)
* Organ transplantation/renal replacement therapy: Prior organ transplant (other than cornea, hair transplant or skin graft), except for history of kidney transplant with subsequent renal failure requiring hemodialysis and for which use of immunosuppressants has been discontinued; Considered for kidney transplant or imminent renal replacement therapy (including intermittent hemodialysis; continuous hemofiltration and hemodialysis; and peritoneal dialysis) for participants with severe renal impairment within a time frame that overlaps with study participation
* Key protocol defined laboratory abnormalities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Sustained Virologic Response at Week 12 After End of Treatment (SVR12) | 12 weeks after end of treatment (EOT) (Week 12 of follow-up phase)
  SVR12 is defined as hepatitis C virus (HCV) ribonucleic acid (RNA) less than (<) lower limit of quantification (LLOQ)
  , detectable or undetectable at 12 weeks after EOT.

SECONDARY OUTCOMES:
Percentage of Participants With On-treatment Response | Baseline up to EOT (Week 12)
  HCV RNA results satisfying a specified threshold. The following thresholds will be considered at any time point: <LLOQ undetectable, <LLOQ detectable, <LLOQ undetectable/detectable.
Percentage of Participants With Sustained Virologic Response at Week 4 After End of Treatment (SVR4) | 4 weeks after EOT (Week 4 of follow-up phase)
  SVR4 is defined as hepatitis C virus (HCV) ribonucleic acid (RNA) less than (<) lower limit of quantification (LLOQ) , detectable or undetectable at 4 weeks after EOT.
Percentage of Participants With Sustained Virologic Response at Week 24 After End of Treatment (SVR24) | 24 weeks after EOT (Week 24 of follow-up phase)
  SVR24 is defined as hepatitis C virus (HCV) ribonucleic acid (RNA) less than (<) lower limit of quantification (LLOQ) , detectable or undetectable at 24 weeks after EOT.
Percentage of Participants With on-treatment Failure | Baseline up to EOT (Week 12), 12 weeks after EOT (Week 12 of follow-up phase)
  Participants who did not achieve SVR12 and with confirmed detectable HCV RNA at the actual end of study treatment.
Percentage of Participants With Viral Relapse | EOT (Week 12) until end of follow-up phase (Week 24 of follow-up phase)
  Participants who did not achieve SVR12, with undetectable HCV RNA at the actual end of study treatment and confirmed HCV RNA >=LLOQ during 24-week follow-up.
Change From Baseline in Hepatitis C Virus (HCV) Nonstructural Protein 3/4A (NS3/4A) and Nonstructural Protein 5A (NS5A) Sequence in Participants not Achieving SVR | Baseline until end of follow-up phase (Week 24 of follow-up phase)
Change From Baseline in HCV Symptom and Impact Questionnaire version 4 (HCV-SIQv4) Overall Body Symptom score | Baseline until end of follow-up phase (Week 24 of follow-up phase)
  The HCV-SIQv4 is a self-administered questionnaire containing 33 items (ranging from 0=Not at All to 4=Extremely): 29 questions developed to assess the severity or frequency of symptoms associated with HCV or its treatment, 3 questions regarding the impact of symptoms on work/school attendance, and 1 question regarding the impact of symptoms on daily activities. Higher HCV-SIQv4 scores indicate worse symptom severity, more time missed from work or school, and more impairment in daily activities, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (6):
- France (3):
  - Paris
  - Toulouse
  - Villejuif
- Spain (3):
  - Barcelona
  - Madrid
  - Santander